CLINICAL TRIAL: NCT01021215
Title: Modulation of Arachidonic Acid Metabolism by Chemopreventive Agents in Smokers
Brief Title: Zileuton With or Without Celecoxib As Chemopreventive Agents in Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2013-00730; NCI-2013-00730 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0804 (Other: M D Anderson Cancer Center); 2009-0804 (Other: DCP); N01CN35159 (NIH)
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2013-10

CONDITIONS: Tobacco Use Disorder
Keywords: Cancer Prevention; Smoking-related lung disease; Smoking; Celecoxib; Celebrex; Zileuton; Zyflo CR; Prevention
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — zileuton; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: Zileuton (Experimental): Zileuton 1200 mg twice orally twice a day on days 1-6.
  Interventions: Drug: Zileuton; Other: laboratory biomarker analysis
- Arm II: Zileuton and Celecoxib (Experimental): Combined Zileuton 1200 mg twice daily plus Celecoxib 200 mg twice daily on days 1-6.
  Interventions: Drug: Zileuton; Drug: Celecoxib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Zileuton — 1200 mg twice daily given orally (PO) for 6 days
  Other Names: Zyflo CR
Drug: Celecoxib — 200 mg twice daily given orally for 6 days
  Other Names: Celebrex
  Arms: Arm II: Zileuton and Celecoxib
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The goal of this clinical research study is to learn how zileuton alone or the combination of zileuton and celecoxib may affect certain chemicals in the body that may be linked with a risk for smoking-related lung disease. These effects will be measured by a urine test

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether short-term administration of zileuton, a 5-lipoxygenase (5-LO) inhibitor, in current smokers will suppress the formation of urinary leukotriene E4 (LTE4) and shunt arachidonic acid into the cyclooxygenase (COX) pathway, resulting in elevated urinary prostaglandin E-metabolite (PGE-M).

SECONDARY OBJECTIVES:

I. To determine whether short-term co-administration of celecoxib, a selective COX-2 inhibitor, and zileuton suppresses levels of both urinary LTE4 and PGE-M in current smokers.

II. To evaluate the association between baseline levels of urinary LTE4 and magnitude of the arachidonic acid shunt induced by zileuton.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive zileuton orally (PO) twice daily (BID) on days 1-6.

ARM II: Patients receive zileuton as in Arm I and celecoxib PO BID on days 1-6.

ELIGIBILITY:
Inclusion Criteria:

* Male or female current tobacco smokers with more or equal to 10 pack years of self-reported smoking exposure and an average of more or equal to 10 cigarettes/day
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky 70-100%)
* Total bilirubin less or equal to 2 * upper limit of normal (ULN)
* Direct bilirubin less or equal to 2 * ULN
* aspartate aminotransferase (AST)/(SGOT) less or equal to 2 * ULN
* alanine aminotransferase (ALT)/(SGPT) less or equal to 2 * ULN
* Alkaline phosphatase less or equal to 2 * ULN
* If the participant is female, of childbearing potential and not lactating, she has a documented negative serum pregnancy test within 14 days prior to randomization

Exclusion Criteria:

* The participant has active cancer (excluding non-melanoma skin cancer)
* The participant has a history of curatively treated cancer with surgical therapy finished within 6 months prior to the Screening visit; or has had chemotherapy, cancer-related immunotherapy, hormonal therapy (other than Hormone replacement therapy (HRT) for menopause), or radiation therapy within 12 months of the screening visit
* The participant has a chronic inflammatory condition, including but not limited to, ulcerative colitis, Crohn's disease, rheumatoid arthritis, psoriasis, gout and pancreatitis
* The participant has an ongoing or active infection, including but not limited to HIV, pneumonia, urinary tract infection
* The participant has a history of nonsteroidal anti-inflammatory drugs (NSAIDs) use, including aspirin (low-dose aspirin also prohibited) and selective COX-2 inhibitors within the previous 4 weeks
* The participant has used zileuton or a leukotriene receptor antagonist within the previous 4 weeks
* The participant has a history of corticosteroid use (excluding topical nasal sprays and dermal application) within the last 6 weeks
* The participant has an acute or chronic kidney disorder
* The participant exhibits clinical evidence of active liver disease or history of chronic liver disease
* The participant has active cardiac disease, or a history of myocardial infarction, angina or coronary artery disease within the past 6 months
* The participant has a history of a cerebrovascular accident (CVA) or transient ischemic attack (TIA)
* The participant has a bleeding history
* The participant is taking drugs known to interact with zileuton or celecoxib, including theophylline, warfarin, propranolol, fluconazole or lithium
* The participant has received any investigational medication within 30 days of the screening visit or is scheduled to receive an investigational agent during the study
* The participant is pregnant or nursing; women must not be pregnant or lactating
* The participant is a female of child-bearing potential (women are considered not of childbearing potential if they are at least two years postmenopausal and/or surgically sterile) who has not used adequate contraception (abstinence; barrier methods such as intrauterine device (IUD), diaphragm with spermicidal gel, condom, or others; and hormonal methods such as birth control pills or others) since her last menses prior to study entry
* The participant is a female of child-bearing potential or male who does not agree to use adequate contraception for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* The participant has participated in the study previously and was withdrawn
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing participants or those who are HIV-positive will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Powel Brown, MD, Principal Investigator — University of Texas (UT) MD Anderson Cancer Center
Locations (2):
- United States (2):
  - Weill Cornell Medical College in New York City, Cornell University, New York, New York
  - MD Anderson Cancer Center - Consortium Lead Organzation, Houston, Texas

REFERENCES:
- See also: University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 5, 2010 to September 12, 2011. All recruitment done in medical clinics at Weill Cornell Medical College (WCMC), a Participating Organization within the MD Anderson Cancer Center (MDACC) Consortium.
Pre-assignment Details: A total of 84 subjects were enrolled, four withdrew for different reasons before beginning study medication leaving 80 subjects started on the study medication(s).
Period: Overall Study
Arm/Group | Arm I: Zileuton | Arm II: Zileuton and Celecoxib
Started | 60 | 20
Received Allocated Intervention | 60 | 20
Completed | 57 | 20
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Of the 80 participants treated three (3) were lost to follow up leaving 77 who completed treatment, and of those reflected as a subset are the 70 compliant participants who completed treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Zileuton | Arm II: Zileuton and Celecoxib | Total
Number analyzed (Participants) | 60 | 20 | 80
Age, Continuous [Median (Full Range); unit: years] | 45 [25 to 64] | 43 [30 to 54] | 43 [25 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 32
  Male | 36 | 12 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 7 | 35
  White | 31 | 10 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 60 | 20 | 80
Smoking (Packs per Year) [Median (Full Range); unit: cigarette packs] — Number of cigarette packs smoked annually; Measure includes the 70 compliant participants only.
  cigarette packs | 19.5 [10 to 68] | 19.5 [10 to 40] | 19.5 [10 to 68]
Baseline PGE-M (ng/mg Cr) [Median (Full Range); unit: ng/mg Cr] — Prostaglandin E metabolite (PGE-M) levels via creatinine (Cr) in the urine measured by a chemical assay. Baseline measure includes the 70 compliant study participants only.
  ng/mg Cr | 12.8 [1.4 to 50.4] | 10.2 [2.3 to 35.1] | 12.6 [1.4 to 50.4]
Baseline LTE4 (pg/mg CR) [Median (Full Range); unit: pg/mg CR] — Leukotriene E4 (LTE4) levels via creatinine (Cr) in the urine measured by a chemical assay. Baseline measure includes the 70 compliant study participants only.
  pg/mg CR | 107 [4 to 268] | 86.5 [37 to 250] | 102.5 [4 to 268]
Gender, Male/Female: Compliant Participants [Number; unit: participants] — Measure includes the 70 compliant study participants only.
  participants
    Female | 19 | 8 | 27
    Male | 33 | 10 | 43
Race, Compliant Participants [Number; unit: participants] — Baseline measure includes the 70 compliant study participants only.
  participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 28 | 7 | 35
    White | 24 | 9 | 33
    Unknown or Not Reported | 0 | 0 | 0
Age, Continuous, Compliant Participants [Mean (Standard Deviation); unit: years] — Baseline measure includes the 70 compliant study participants only.
  years | 43.8 (9.6) | 43.1 (7.6) | 43.6 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Median Urinary PGE-M Levels (Pre and Post Treatment)
Description: Pre and Post treatment differences in urinary PGE-M levels measured in each treatment arm. PGE-M levels reported as median with full range (ng/mg creatinine) for Pre treatment versus Post treatment PGE-M levels among study participants compliant to treatment with evaluable urine samples at both time points (baseline and Day 6 +/- 1 day).
Time Frame: Baseline and Day 6
Population: Seventy-seven subjects completed the entire study with seven of those excluded from analysis as non-compliant (study medications were undetectable). Urine of two participants contained interfering substances thus were excluded from PGE-M related analysis.
Measure: Median (Full Range); unit: ng/mg creatinine
Arm/Group | Arm I: Zileuton | Arm II: Zileuton and Celecoxib
Number analyzed (Participants) | 52 | 16
ng/mg creatinine
  Pre PGE-M Levels | 12.8 [1.4 to 50.4] | 13.4 [2.3 to 35.1]
  Post PGE-M Levels | 10.5 [2.0 to 34.6] | 3.9 [1.2 to 10.1]

2. Primary Outcome: Median Urinary LTE4 Levels (Pre and Post Treatment)
Description: Pre and Post treatment differences in urinary LTE4 levels measured in each treatment arm compared using paired t-test should the data conform to the normality assumption or one-sample Wilcoxon rank-sum test. LTE4 levels reported as median with full range (pg/mg creatinine) for Pre treatment versus Post treatment LTE4 levels among study participants compliant to treatment with evaluable urine samples at both time points (baseline and Day 6 +/- 1 day).
Time Frame: Baseline and day 6
Population: Seventy-seven subjects completed the entire study, three withdrew for personal reasons. Seven of those participants were excluded from analysis as non-compliant (study medications were undetectable).
Measure: Median (Full Range); unit: pg/mg creatinine
Arm/Group | Arm I: Zileuton | Arm II: Zileuton and Celecoxib
Number analyzed (Participants) | 52 | 18
pg/mg creatinine
  Pre LTE4 levels | 107 [4 to 268] | 86 [37 to 250]
  Post LTE4 levels | 42 [4 to 292] | 30 [10 to 84]

3. Secondary Outcome: Proportion of Cases With a Post-treatment Increase in Urinary PGE-M Levels
Description: Proportion of cases with a post-treatment increase in urinary PGE-M levels by comparing those treated with Zileuton and Celecoxib combined therapy compared to those treated with Zileuton alone. Pre/postchange in levels (Increase) derived from baseline level to Day 6 +/- 1 day. Differences in baseline levels between 2 treatment arms were examined using the Wilcoxon rank-sum test.
Time Frame: Baseline to Day 6
Population: Analysis includes only number of participants in each treatment arm with post-treatment increase in urinary PGE-M levels as measured from baseline.
Measure: Number; unit: proportion of participants
Arm/Group | Arm I: Zileuton | Arm II: Zileuton and Celecoxib
Number analyzed (Participants) | 52 | 16
proportion of participants | .37 | .06

ADVERSE EVENTS:
Time Frame: All adverse events that occur after the informed consent signed (including run-in) until subject off study. Study period was from May 2010 to September 2011.
Description: Common Toxicity reporting for the study began with Common Toxicity Criteria for Adverse Effects (CTCAE) version 3.0 and completed with CTCAE version 4.0. Reporting has been combined in the provided tables.
Arm/Group | Arm I: Zileuton | Arm II: Zileuton and Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/20
Other Adverse Events (participants affected / at risk) | 26/60 | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Zileuton (N=60) | Arm II: Zileuton and Celecoxib (N=20)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0
DIARRHEA (Gastrointestinal disorders) | 5 | 0
DIZZINESS (Nervous system disorders) | 3 | 0
DRY MOUTH (Gastrointestinal disorders) | 3 | 1
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0
EYE PAIN (Eye disorders) | 1 | 0
FATIGUE (General disorders) | 4 | 1
FLATULENCE (Gastrointestinal disorders) | 2 | 0
GERD (Gastrointestinal disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 5 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0
IRRITABILITY (General disorders) | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 2
PAIN IN EXTREMITY (Vascular disorders) | 1 | 0
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RESTLESSNESS (Psychiatric disorders) | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 | 0
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 | 1
WATERING EYES (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less